CLINICAL TRIAL: NCT07334652
Title: Pain and Comfort in the Examination of Retinopathy of Prematurity
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Türkan Kadiroğlu, Associate Professor, PhD, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: B.30.2.ATA.0.01.00/648; Ataturk University (Other: Scientific Research Projects Coordination Centre)
Record Dates: First submitted 2025-12-31; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Premature; Retinopaty of Prematurity
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pacifier group (Experimental): Breast milk and dummy
  Interventions: Other: Pacifier group
- Control Group (No Intervention): Routıne Procedure

INTERVENTIONS:
Other: Pacifier group — During the examination, babies will be given a dummy dipped in breast milk.
  Arms: Pacifier group

SUMMARY:
This study is planned to be conducted in the Neonatal Intensive Care Unit using a double-blind, parallel-group, randomised controlled design to determine the effect of a pacifier dipped in breast milk on pain and comfort during Retinopathy of Prematurity examinations. The study will be conducted in the Neonatal Intensive Care Unit of a University Hospital in Erzurum. The sample for the study will consist of preterm infants born before 32 weeks of gestation who are receiving treatment and care at the clinic during the study period and who meet the study criteria, without using any sampling method. The power analysis for sample size indicated that at least 36 infants should be included in the study, with 18 infants in each of the experimental and control groups. The control group will undergo ROP examination in accordance with standard clinical procedures. All examinations will be performed by the same ophthalmologist. Infants in the experimental group will be fed with a pacifier dipped in breast milk, starting two minutes prior to the examination, by the same clinical nurse responsible for the infant's care, and feeding will continue until the examination is completed. Video recordings will be taken of all infants from two minutes prior to the start of the examination until two minutes after the examination. In both groups, data will be monitored and recorded using the Preterm Infant Pain Profile-Revised (PIPP-R), the Preterm Infant Comfort Scale (COMFORT neo), and vital signs before the ROP examination begins, during the examination, and after the examination.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age ≤ 32 weeks
* Birth weight ≤ 2000 grams
* Infants undergoing their first ROP examination
* Spontaneous breathing, not intubated,
* Not receiving sedation
* No congenital defects,
* No unexplained crying,
* No surgical intervention,
* Parents' consent to participate in the study

Exclusion Criteria:

* The presence of a condition that prevents pain assessment (intracranial haemorrhage, neurodevelopmental delay, etc.)
* A different painful procedure performed prior to ROP (one hour)
* Being on mechanical ventilation
* Administration of sedative, analgesic, and anticonvulsant medication prior to examination

Ages: 0 Months to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Procedural pain | 8-12 week
  Premature Infant Pain Profile - Revision (PIPP-R)

SECONDARY OUTCOMES:
Comfort | 8-12 week
  Preterm infant comfort scale (COMFORT neo)

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University Faculty of Nursing, Erzurum, Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No